CLINICAL TRIAL: NCT03038633
Title: A Trial to Evaluate the Safety and Tolerability of a Novel Medical Food for Management of Iron Deficiency Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey J. Pu, MD, PhD, Assistant Proffesor of Medicine, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 34696
Record Dates: First submitted 2015-10-27; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Individuals will receive 300 mg capsules of the novel medical food. The iron content of these capsules is 7.4mg. Our initial dose is set at 22.2 mg of iron. This dose was chosen as the initial starting dose because it is within the range of the RDA for iron for adult women (18mg). Thus this dose is considered the minimum that would be utilized in any setting for maintenance of a healthy iron status. The dosing increases to a maximum of 88.8mg of iron per day which is significantly below the standard amount of iron (165-195mg per day) recommended for an iron deficient individual or the amount of iron given intravenously (1000 mg) for some iron deficient conditions. As mentioned, the total element iron given a patient treated with FAS is up to 190mg of iron. Assuming a 10% absorption rate these patients get 19mg of iron. So if our goal is approximately 19mg of iron absorbed per day and we assume a 50% absorption rate then our target dose is 6-9 capsules per day (44.4-66.6 mg iron).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 (Experimental): 900 mg novel medical food containing 22.2mg iron
  * receive 900 mg by mouth (3 capsules, one at each meal) daily; after Day 28 remain on level for additional 2 months if clinically indicated
  * receive a phone call from coordinator between Day 5-9 to assess side effects and medications
  * return to General Clinical Research Center, (GCRC) for a blood draw at days 14, 28, 60, and 90 while on novel medical food
  Interventions: Other: Novel Medical Food
- Cohort 2 (Experimental): 1800 mg novel medical food containing 44.4 mg of iron
  * receive 1800 mg by mouth (3 capsules, one at each meal) daily; after Day 28 remain on level for additional 2 months if clinically indicated
  * receive a phone call from coordinator between Day 5-9 to assess side effects and medications
  * return to GCRC for a blood draw at days 14, 28, 60, and 90 while on novel medical food
  Interventions: Other: Novel Medical Food
- Cohort 3 (Experimental): 2700 mg novel medical food containing 66.6 mg of iron
  * receive 2700 mg by mouth (3 capsules, one at each meal) daily; after Day 28 remain on level for additional 2 months if clinically indicated
  * receive a phone call from coordinator between Day 5-9 to assess side effects and medications
  * return to GCRC for a blood draw at days 14, 28, 60, and 90 while on novel medical food
  Interventions: Other: Novel Medical Food
- Cohort 4 (Experimental): 3600 mg novel medical food containing 88.8 mg of iron
  * receive 3600 mg by mouth (3 capsules, one at each meal) daily; after Day 28 remain on level for additional 2 months if clinically indicated
  * receive a phone call from coordinator between Day 5-9 to assess side effects and medications
  * return to GCRC for a blood draw at days 14, 28, 60, and 90 while on novel medical food
  Interventions: Other: Novel Medical Food

INTERVENTIONS:
Other: Novel Medical Food — This medical food takes advantage of the stability and high level of solubility of the human H-ferritin protein to be absorbed by the body as an iron source; indeed H-ferritin is enriched in breast milk as the mechanism for transferring iron from mother to infants. Once the ferritin has been absorbed from the gut, uptake into each organ is regulated by a specific extracellular receptor pathway to deliver iron in the body's preferred bioavailable form.

SUMMARY:
This is a Phase 1 clinical trial designed to evaluate the safety and tolerability of a novel medical food utilizing a nutritional strain of yeast for management of Iron Deficiency Anemia.

DETAILED DESCRIPTION:
The investigational product is a medical food and is the result of discoveries following extensive research on two preclinical models carried out by a team of researchers at Penn State University. This study will utilize the standard "3+3" rule-based dose-escalation schemes, which use predetermined dose levels and cohorts of three patients. The total time commitment for each subject is approximately three months.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin, (Hgb) 7-10 g/dL; transferrin saturation <20%; and serum ferritin <20ng/mL

Exclusion Criteria:

* Pregnant or sexually-active female subjects who are of childbearing potential and who are not willing to use an acceptable form of contraception (tubal ligation or otherwise be incapable of pregnancy, hormonal contraceptives, spermicide plus barrier or intrauterine device).
* Present consumption of iron supplements or multivitamins must be switched to vitamins not containing iron, such as the multivitamin Centrum Silver. No washout period is necessary since it will be apparent from the ongoing anemia that any current supplements are ineffective.
* Current anemia not attributed to immune deficiency, (ID) (e.g. other microcytic anemia or hemolytic, macrocytic, sideroblastic or myelosuppression or chemotherapy or radiotherapy induced anemia).
* Active malignancy within 1 year. Basal or squamous cell skin cancer is not exclusionary.
* Aspartate Aminotransferase, (AST) or Alanine Aminotransferase, (ALT) at screening greater than 1.5 times the upper limit of normal.
* Known positive hepatitis B with evidence of active hepatitis.
* Known positive HIV-1/HIV-2 antibodies (anti-HIV).
* Patient has a current diagnosis of asthma and is actively using an anti-asthmatic therapy.
* Received an investigational drug within 30 days of screening.
* Hemochromatosis or other iron storage disorders.
* Unregulated hypertension
* Chronic kidney disease.
* Chronic inflammatory condition including but not limited to Lupus and Rheumatoid Arthritis.
* Significant cardiovascular disease, including but not limited to myocardial infarction or unstable angina within 6 months prior to study inclusion or current history of New York Heart Association, (NYHA) Class III or IV congestive heart failure.
* Smoking
* Irritable Bowel Syndrome
* Any other laboratory abnormality, medical condition or psychiatric disorder which in the opinion of the investigator puts the subject's disease management at risk or may result in the subject being unable to comply with study requirements.
* Breastfeeding planned on or after enrolling in the study.
* Known allergy to yeast
* Currently on Monoamine oxidase inhibitors, (MAOI's) or Demerol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity, (DLT) | 28 Days
  Still evaluating data

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data under review